CLINICAL TRIAL: NCT04144322
Title: Short Dental Implants (5 mm) Versus Long Dental Implants (10 mm) in Combination With Sinus Floor Elevation: A Randomized Clinical Trial
Brief Title: Short Dental Implants (5 mm) Versus Long Dental Implants (10 mm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Tae-Ju Oh, Clinical Professor of Dentistry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00151047
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Bone Loss, Alveolar
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Short Implant (Other): 17 patients will receive a 5 mm short implant.
  Interventions: Device: Zimmer T3 Short Ex Hex With Discrete Crystalline Deposition
- Long Implant (Other): 17 patients will receive a sinus lift procedure, bone graft, and 10 mm implant.
  Interventions: Device: Zimmer T3 with Discrete Crystalline Deposition Ex Hex Parallel Walled implants

INTERVENTIONS:
Device: Zimmer T3 Short Ex Hex With Discrete Crystalline Deposition — Placement of a short implant
  Arms: Short Implant
Device: Zimmer T3 with Discrete Crystalline Deposition Ex Hex Parallel Walled implants — Placement of a long implant with sinus lift and bone graft
  Arms: Long Implant

SUMMARY:
The purpose of this study is to evaluate the survival rate of 5 mm short implants compared to longer implants (10 mm) placed in sinus-grafted sites.

Primary aim: Compare bone loss between the two groups Secondary aim: Compare surgical time and patient-reported outcomes (satisfaction and post-operative pain)

DETAILED DESCRIPTION:
34 patients requiring an implant to replace an upper missing tooth in the premolar or 1st molar area with a bone crest height from 5 to 8 mm will be recruited for this trial. Patients will be randomized to either the test (5-mm implant) or control group (10-mm implant) using a computer-generated randomization list . 17 patients will receive a sinus lift procedure, bone graft, and 10 mm implant while the other 17 patients will receive a 5 mm short implant.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70 years at enrollment
* Systemically healthy patients
* Full-mouth plaque score and full-mouth bleeding score ≤ 30% (measured at four sites per tooth)
* In need of one premolar or 1st molar dental implant in the maxillary area
* Neighboring teeth to the planned implant must have natural root(s) or implant supported restoration.
* Presence of natural tooth/teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned crown/s deemed by the investigator as likely to present an initially stable implant situation
* Residual bone height under the maxillary sinus between 5 to 7 mm and a width of at least 7 mm, as measured on cone beam computer tomography (CBCT) scans.

Exclusion Criteria:

* Unlikely to be able to comply with study procedures
* Uncontrolled pathologic processes in the oral cavity
* History of head and neck chemotherapy within 5 years prior to surgery
* Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration
* Uncontrolled diabetes mellitus HbA1c >8
* Taking corticosteroids, IV bisphosphonates, or any other medication that could influence post-operative healing and/or osseointegration
* Smokes more than 10 cigarettes/day
* Bruxer
* Present alcohol and/or drug abuser
* Pregnant, unsure pregnancy status, or lactating females (self-reported)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Ju Oh, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anitua E, Alkhraist MH, Pinas L, Begona L, Orive G. Implant survival and crestal bone loss around extra-short implants supporting a fixed denture: the effect of crown height space, crown-to-implant ratio, and offset placement of the prosthesis. Int J Oral Maxillofac Implants. 2014 May-Jun;29(3):682-9. doi: 10.11607/jomi.3404. PMID 24818208
- [Background] Anitua E, Pinas L, Orive G. Retrospective study of short and extra-short implants placed in posterior regions: influence of crown-to-implant ratio on marginal bone loss. Clin Implant Dent Relat Res. 2015 Feb;17(1):102-10. doi: 10.1111/cid.12073. Epub 2013 May 8. PMID 23656303
- [Background] Buser D, Janner SF, Wittneben JG, Bragger U, Ramseier CA, Salvi GE. 10-year survival and success rates of 511 titanium implants with a sandblasted and acid-etched surface: a retrospective study in 303 partially edentulous patients. Clin Implant Dent Relat Res. 2012 Dec;14(6):839-51. doi: 10.1111/j.1708-8208.2012.00456.x. PMID 22897683
- [Background] Sargozaie N, Moeintaghavi A, Shojaie H. Comparing the Quality of Life of Patients Requesting Dental Implants Before and After Implant. Open Dent J. 2017 Aug 31;11:485-491. doi: 10.2174/1874210601711010485. eCollection 2017. PMID 29114333
- [Background] Pieri F, Forlivesi C, Caselli E, Corinaldesi G. Short implants (6mm) vs. vertical bone augmentation and standard-length implants (>/=9mm) in atrophic posterior mandibles: a 5-year retrospective study. Int J Oral Maxillofac Surg. 2017 Dec;46(12):1607-1614. doi: 10.1016/j.ijom.2017.07.005. Epub 2017 Jul 24. PMID 28751181
- [Background] Lemos CA, Ferro-Alves ML, Okamoto R, Mendonca MR, Pellizzer EP. Short dental implants versus standard dental implants placed in the posterior jaws: A systematic review and meta-analysis. J Dent. 2016 Apr;47:8-17. doi: 10.1016/j.jdent.2016.01.005. Epub 2016 Jan 19. PMID 26804969
- [Background] Garaicoa-Pazmino C, Suarez-Lopez del Amo F, Monje A, Catena A, Ortega-Oller I, Galindo-Moreno P, Wang HL. Influence of crown/implant ratio on marginal bone loss: a systematic review. J Periodontol. 2014 Sep;85(9):1214-21. doi: 10.1902/jop.2014.130615. Epub 2014 Jan 20. PMID 24444399
- [Background] Fan T, Li Y, Deng WW, Wu T, Zhang W. Short Implants (5 to 8 mm) Versus Longer Implants (>8 mm) with Sinus Lifting in Atrophic Posterior Maxilla: A Meta-Analysis of RCTs. Clin Implant Dent Relat Res. 2017 Feb;19(1):207-215. doi: 10.1111/cid.12432. Epub 2016 Jun 13. PMID 27295262
- [Background] Chappuis V, Araujo MG, Buser D. Clinical relevance of dimensional bone and soft tissue alterations post-extraction in esthetic sites. Periodontol 2000. 2017 Feb;73(1):73-83. doi: 10.1111/prd.12167. PMID 28000281
- [Background] Schneider CA, Rasband WS, Eliceiri KW. NIH Image to ImageJ: 25 years of image analysis. Nat Methods. 2012 Jul;9(7):671-5. doi: 10.1038/nmeth.2089. PMID 22930834
- [Background] Strietzel FP, Reichart PA. Oral rehabilitation using Camlog screw-cylinder implants with a particle-blasted and acid-etched microstructured surface. Results from a prospective study with special consideration of short implants. Clin Oral Implants Res. 2007 Oct;18(5):591-600. doi: 10.1111/j.1600-0501.2007.01375.x. Epub 2007 Jun 21. PMID 17590161
- [Background] Telleman G, Raghoebar GM, Vissink A, Meijer HJ. Impact of platform switching on peri-implant bone remodeling around short implants in the posterior region, 1-year results from a split-mouth clinical trial. Clin Implant Dent Relat Res. 2014 Feb;16(1):70-80. doi: 10.1111/j.1708-8208.2012.00461.x. Epub 2012 May 11. PMID 22577959
- [Background] Thoma DS, Haas R, Sporniak-Tutak K, Garcia A, Taylor TD, Hammerle CHF. Randomized controlled multicentre study comparing short dental implants (6 mm) versus longer dental implants (11-15 mm) in combination with sinus floor elevation procedures: 5-Year data. J Clin Periodontol. 2018 Dec;45(12):1465-1474. doi: 10.1111/jcpe.13025. Epub 2018 Nov 25. PMID 30341961

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Short Implant | Long Implant
Started | 17 | 17
Completed | 15 | 15
Not Completed | 2 | 2
Not completed — Lack of Efficacy | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Implant | Long Implant | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.67 (14.57) | 56.87 (13.31) | 57.76 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 5 | 9 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Soft tissue phenotype [Count of Participants; unit: Participants]
  Thin | 1 | 3 | 4
  Medium | 5 | 7 | 12
  Thick | 3 | 2 | 5
  Very Thick | 6 | 3 | 9
Bone density [Count of Participants; unit: Participants] — Subjective evaluation of the bone type (Lekholm & Zarb 1985) during implant site preparation performed by the surgeon.
  * D1: Almost entirely comprised of homogeneous compact bone (most dense)
  * D2: thick layer of compact bone surrounding a core of dense trabecular bone
  * D3: thin layer of cortical bone surrounding a core of dense trabecular bone
  * D4: Thin layer of cortical bone surrounding a core of low-density trabecular bone coupled with the surgeon's tactile perception (least dense)
  Participants
    D1 | 0 | 0 | 0
    D2 | 0 | 2 | 2
    D3 | 15 | 13 | 28
    D4 | 0 | 0 | 0
Residual ridge height [Mean (Standard Deviation); unit: millimeters] | 5.74 (0.84) | 6.39 (1.53) | 6.07 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mesial-distal (M-D) Bone Loss
Description: Comparing mesial-distal (M-D) bone loss between the two groups. This will be measured in millimeters using standardized radiographs of the implant site at the screening visit, surgical visit, 4 months post-op, 5 months post-op, 12 months post-op, and 24 months post-op visits.
Time Frame: Baseline, surgical visit 1 day, 4 months, 5 months, 12 months, 24 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Short Implant | Long Implant
Number analyzed (Participants) | 15 | 15
millimeters
  Surgery visit | 0.63 (0.38) | 0.61 (0.57)
  4 months (second stage) | -0.41 (0.76) | -0.40 (1.04)
  5 months (loading) | -0.55 (0.83) | -0.64 (0.75)
  12 months | -0.74 (0.79) | -0.40 (0.57)
  24 months | -0.84 (0.62) | -059 (0.65)

2. Secondary Outcome: Survival Rate
Description: The survival rate of the two groups will be recorded as a percentage at the 5 month post-op, 12 month post-op, and 24 month post-op visits based on clinician assessment.
Time Frame: 5 month post-op, 12 month post-op, and 24 month post-op visits
Measure: Count of Participants; unit: Participants
Arm/Group | Short Implant | Long Implant
Number analyzed (Participants) | 17 | 17
Participants
  5 months (loading) | 17 | 15
  12 months | 17 | 15
  24 months | 15 | 15

3. Secondary Outcome: Number of Sites With Bleeding on Probing
Description: The number of sites with bleeding on probing will be compared between the two groups. Bleeding on probing of the implant site will be measured with a periodontal probe at the 5 month post-op, 12 month post-op, and 24 month post-op visits.
Time Frame: 5 month post-op, 12 month post-op, and 24 month post-op visits
Measure: Mean (Standard Deviation); unit: implant sites
Arm/Group | Short Implant | Long Implant
Number analyzed (Participants) | 15 | 15
implant sites
  5 months (loading) | .03 (.02) | .08 (.05)
  12 months | .14 (.05) | .39 (.09)
  24 months | .35 (.07) | .32 (.08)

4. Secondary Outcome: Probing Pocket Depth
Description: The probing pocket depths will be compared between the two groups. Probing depths of the implant site will be measured with a periodontal probe at the 5 month post-op, 12 month post-op, and 24 month post-op visits.
Time Frame: 5 month post-op, 12 month post-op, and 24 month post-op visits
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Short Implant | Long Implant
Number analyzed (Participants) | 15 | 15
millimeters
  5 months (loading) | 2.84 (0.15) | 2.94 (.15)
  12 months | 3.32 (0.14) | 3.27 (.15)
  24 months | 3.79 (0.16) | 3.72 (.16)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during each subject's entire participation in the study (approximately 2 years)
Arm/Group | Short Implant | Long Implant
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/17 | 3/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Implant (N=17) | Long Implant (N=17)
Appendicitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Subject noted having some gastrointestinal discomfort earlier that week before their baseline surgery. The next day, the subject notified one of the co-investigators that they had to go to the hospital for emergency surgery to remove their appendix.
Coronavirus disease of 2019 and ablation (Cardiac disorders) | 0 (0) | 1 (1) — Subject contracted coronavirus disease of 2019 and was hospitalized for 10 days, then later needed to have a heart ablation.
Vehicle accident (Social circumstances) | 2 (2) | 0 (0) — Severe vehicle accident that required hospitalization.
Assault (Social circumstances) | 0 (0) | 1 (1) — Physically assaulted by someone which required physical therapy for many months.
Hip replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT04144322/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT04144322/ICF_001.pdf